CLINICAL TRIAL: NCT03422796
Title: The Effect of Sumatriptan and Placebo Injection on Cilostazol Induced Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Katrine Falkenberg, Medical doctor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-17026731
Record Dates: First submitted 2017-10-20; First posted 2018-02-06 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Cilostazol; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sumatriptan (Active Comparator): headache is induced with Cilostazol. This headache is treated double-blinded with 6mg/ml sumatriptan
  Interventions: Drug: Cilostazol 200mg; Drug: SUMAtriptan 6 MG/ML
- Placebo (Placebo Comparator): headache is induced with Cilostazol. This headache is treated double-blinded with 1 tablet of placeb
  Interventions: Drug: Cilostazol 200mg; Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol 200mg — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Pletal
Drug: SUMAtriptan 6 MG/ML — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Imigran
  Arms: Sumatriptan
Drug: Placebo — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Arms: Placebo

SUMMARY:
To develop a pragmatic migraine model the investigators will induce headache in patients with migraine without aura with a phosphodiesterase inhibitor (cilostazol). If the headache responds to sumatriptan injection, the model can be used to test new drug candidates.

DETAILED DESCRIPTION:
There remains a great need for more effective anti-migraine drugs with fewer side effects. Human experimental models are valuable in early phase development of new anti-migraine drugs but useful models have not yet been developed. The investigators' group has shown that Cilostazol, a phosphodiesterase inhibitor induce headache/migraine in both healthy volunteers and in patients with migraine without aura (MO). To validate this model, the headache must respond to specific migraine treatment with sumatriptan.

Hypothesis: Cilostazol induces a migraine-like headache in MO-patients and the induced headache responds to sumatriptan injection Aim: Developing a pragmatic and valid model for the testing of new anti-migraine drugs.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients who meet IHS criteria for migraine with or without aura of both sexes
* 18-70 years
* 45-95 kg.

Exclusion Criteria:

* Any other type of headache then migraine without aura (except episodic tension-type headache < 1 day per week)
* Serious somatic or psychiatric disease
* Pregnancy
* Intake of daily medication (except oral contraceptives)
* Triptan non-responders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Difference in median headache score after sumatriptan/placebo | 2hours
  The investigators will assess the outcome measures 1 year after the beginning of the study
difference in AUC 0-4h post treatment | 4hours
  The difference in area under the curve 0-4h after treatment with sumatriptan and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falkenberg K, Bjerg HR, Olesen J. Subcutaneous sumatriptan reduces cilostazol induced headache in migraine patients. Cephalalgia. 2020 Jul;40(8):842-850. doi: 10.1177/0333102420915166. Epub 2020 Mar 26. PMID 32216457